CLINICAL TRIAL: NCT05769101
Title: Effects of a Protein-Based Multi-Ingredient Recovery Supplement Combined With Resistance Training on Body Composition, Performance, Muscular Properties, and Wellbeing on Middle-Aged and Older Adults.
Brief Title: Effects of a Recovery Supplement on Body Composition, Performance, Muscular Properties, and Wellbeing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Joel Puente (Other)
Collaborators: Crown Sport Nutrition (Industry); Go Fit Spain (Unknown)
Responsible Party: Sponsor-Investigator, Joel Puente, Principal Investigator, University of Greenwich
Organization: University of Greenwich (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UGreenwich4
Record Dates: First submitted 2023-02-20; First posted 2023-03-15 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2023-03

CONDITIONS: Protein Deficiency; Training Group, Sensitivity; Fatigue; Muscular Atrophy; Psychological
Keywords: Fatigue; Supplement; Protein; Creatine; Resistance Training; Recovery; Strength; Rate of Perceived Exertion; Muscle
MeSH Terms: conditions — Protein Deficiency; Hypersensitivity; Fatigue; Muscular Atrophy

STUDY DESIGN:
Intervention Model Description: 6 Weeks of resistance training (alternate days), with a post-workout or Maltodextrin intake.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multi-Ingredient Post-Workout Supplement (Experimental): A 60 g dose of a commercially available Recovery supplement providing ~205 kcal including Proteins (+EAA), Carbohydrates, Creatine, and Vitamin D. Diluted in 350 ml of water.
  Interventions: Dietary Supplement: Ingestion of a Post-Workout Supplement
- Maltodextrin Supplement (Placebo Comparator): An isoenergetic Maltodextrin supplement will be administered as placebo. Dissolved in 350 ml of water.
  Interventions: Dietary Supplement: Ingestion of a Maltodextrin Supplement

INTERVENTIONS:
Dietary Supplement: Ingestion of a Post-Workout Supplement — The Post-Workout Supplement is administered 15 minutes after the completion of training sessions. No supplementation is administered in non-training days. The Resistance Training is performed in alternate days. The training Protocol is: 10 minutes of standardized warm-up, Strength Circuit training using free weights (Alternate Box Step-Ups, Bench Press; Parallel Squat; Up-right Row; Deadlift; Alternate Lunges; Shoulder Press; Leg Extension). The participants perform 16 repetitions of each exercise, with 30 seconds rest and 3 minutes rest after every set. If they can complete 16 repetitions easily, 2.5 to 5 kg are added for the next set. Also, whole-body Perceptual Response is assessed using the 0-10 OMNI-RES Scale, after every set and 15 minutes after finishing.
  Arms: Multi-Ingredient Post-Workout Supplement
Dietary Supplement: Ingestion of a Maltodextrin Supplement — The Maltodextrin Supplement is administered 15 minutes after the completion of training sessions. No supplementation is administered in non-training days. The Resistance Training is performed in alternate days. The training Protocol is: 10 minutes of standardized warm-up, Strength Circuit training using free weights (Alternate Box Step-Ups, Bench Press; Parallel Squat; Up-right Row; Deadlift; Alternate Lunges; Shoulder Press; Leg Extension). The participants perform 16 repetitions of each exercise, with 30 seconds rest and 3 minutes rest after every set. If they can complete 16 repetitions easily, 2.5 to 5 kg are added for the next set. Also, whole-body Perceptual Response is assessed using the 0-10 OMNI-RES Scale, after every set and 15 minutes after finishing.
  Arms: Maltodextrin Supplement

SUMMARY:
The investigation will be conducted as a double blinded, randomized, parallel between treatment conditions comparison design with two different groups ingesting a different supplement each one.

DETAILED DESCRIPTION:
Following inclusion, familiarization and baseline assessments, the participants will be randomly allocated to receive either a multi-ingredient, post-workout supplement (REC) or maltodextrin (CHO). Thereafter, the participants will follow a 6-weeks resistance training mesocycle, involving three resistance training sessions (Monday, Wednesday and Friday) per week (18 sessions in total). Before and after the 6 weeks of intervention, the following assessments will be performed: (i) Body composition (fat mass and fat-free mass) via air displacement plethysmography (BodPod); (ii) muscle contractile properties on Vastus Medialis and Anterior Deltoids (via Tensiomyography; (iii) muscle structure of the Vastus Lateralis of the Quadriceps and the Elbow Flexors of dominant extremities via Ultrasound; (iv) Maximal Isometric Strength (Isometric Mid-Thigh Pull); (v) Upper and Lower Body Muscular Power (Medicine Ball Throw and Vertical Jump), (vi) Upper and Lower Muscular Endurance (30- Seconds Sit-to-Stand and 30-Seconds 16RM Bench Press), (vii) Immune System (via HemoCue WBC DIFF System).

The supplements will be ingested immediately (within 15 min) after each training session.

Energy Feeling Questionnaire will be filled immediately before warming up.

In addition, Rate of Perceived Exertion to training will be assessed 15 min after the completion of all workouts.

ELIGIBILITY:
Inclusion Criteria:

* Healthy (no injuries, illnesses or medication intake).
* Between 45 and 65 years old.
* Active and familiarised with Resistance Training.

Exclusion Criteria:

* Unhealthy (illnesses or medication intake) or injured.
* Untrained.
* Young (<45 y.o.) or elderly (>65 y.o.).

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-05-30 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Vertical Jump | Changes from 3 days previous to, and 3 days after the completion of the 6-weeks training program
  Height (measured in centimetres)
Chest Medicine Ball Throw | Changes from 3 days previous to, and 3 days after the completion of the 6-weeks training program
  Distance (measured in centimetres)
Muscle Thickness | Changes from 3 days previous to, and 3 days after the completion of the 6-weeks training program
  Thickness of the Vastus Lateralis and the Elbow Flexors of the dominant limbs
Self Perceived Energy Feeling | [Time Frame: Changes from 3 days previous to, and 3 days after the completion of the 6-weeks training program]
  All participants will fill a short questionnaire (from 1 to 5 points) about their perception of energy before every training. Energy Feeling will be assessed (Evergy level, Fatigue Level, Feeling of Alertness, and Feeling of Focus for the task, valued from 1 = low energy to 5 = high energy).
White Blood Cells count | Changes from 3 days previous to, and 3 days after the completion of the 6-weeks training program
  White blood cell (WBC) count including a five-part differential

CONTACTS AND LOCATIONS:
Locations (1):
- University of Greenwich, Avery Hill Campus, Sparrows Farm. Avery Hill, London., United Kingdom, SE9 2BT, London, Avery Hill, London., United Kingdom

IPD SHARING:
Plan to Share IPD: No